CLINICAL TRIAL: NCT05451459
Title: Fit Families Program: A Multisite Study
Brief Title: Fit Families Multisite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Syracuse University (Other); University of Northern Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-0165; 2022-0165 (Other: UW Madison); A176000 (Other: UW Madison); 3/15/2022 (Other: UW Madison)
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Developmental Disability; Intellectual Disability
MeSH Terms: conditions — Developmental Disabilities; Intellectual Disability | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group will be offered four one-day group workshops (2-3 hours each) covering topics of 1) Sensory Integration, 2) Communication, 3) Physical activity, and 4) Sports. The workshops will be offered online via Zoom and will be video recorded. The intervention group will also receive information (activity booklets via the Fit Families App) and physical education (physical activity)-related equipment, which will be mailed to them. At the end of the workshop parents will be instructed to practice the skills they learned with their child for the next 3 weeks (for at least 3 hrs per week).
  Interventions: Other: 12-week FMS Intervention; Behavioral: Physical Activities & Activity Booklets (via FitFamilies app)
- Wait-list home-based group (Other): The wait-list home-based group will serve as the control group (during intervention). This group will be instructed to continue their typical routines and activities for the duration of the 12-week intervention. At the end of the 12 weeks, they will be asked to complete the post-test surveys (same as questionnaires completed prior to randomization). Their participation in the research will be complete at this time. However, because the intervention has been shown to potentially benefit families, immediately following the post-test, participants in the wait-list home-based group will be offered the chance to complete the home-based intervention program (e.g., receiving the same intervention protocol and materials (physical education equipment and lesson plans/workbook) as described for the intervention group). No data will be collected for research from them during this time.
  Interventions: Behavioral: Physical Activities & Activity Booklets (via FitFamilies app)

INTERVENTIONS:
Other: 12-week FMS Intervention — 4 virtual workshops (2-3 hours each) covering topics of 1) Sensory Integration, 2) Communication, 3) Physical activity, and 4) Sports (during intervention)
  Arms: Intervention Group
Behavioral: Physical Activities & Activity Booklets (via FitFamilies app) — expected to engage in physical activity at least 3 hours per week, virtual workshops provide them with resources to engage in Physical activity

SUMMARY:
The purpose of the study is twofold. First, the investigator wants to identify the effect of a 12-week online fundamental motor skills (FMS) (e.g., throwing, catching, running) intervention on active participation in physical recreation activities as well as a variety of other factors(parental stress, parental self-efficacy, and children's adaptive skills). Second, the investigator also wants to identify patterns, benefits, constraints, and strategies to active participation in physical recreation activities among families of children with developmental disabilities such as autism, down syndrome, etc (post-program) via focus groups interviews (via zoom) with parents. Participants will be randomly assigned to one of two protocols: 1) Intervention group and 2) wait-listed home-based group. Participants in both groups will receive an activity booklet (in the form of an App) and physical education-related activity items (e.g., ball, hoop). The investigator hypothesizes that both the intervention group will improve in all measures from pre to post compared to the wait-list control group. The study team wants to determine if the differences in the intervention group differ significantly or are equitable in terms of gains in all areas.

DETAILED DESCRIPTION:
Prior to participating in the program, interested families will complete an electronic screening questionnaire via Qualtrics (Initial Screening Evaluation) to identify if their family are eligible to participate in this study. On the Initial Screening Evaluation, parents will be asked to report on their children's previous diagnoses, ambulatory ability, significant behavior needs, ability to follow directions, and independent or assisted communication. Parents will need to confirm that their children are ambulatory and are diagnosed with a developmental disability. Children with significant communication needs will still be considered for the study. No new disability diagnostic assessment will be conducted. Diagnostic severity of disability will not be a factor in recruitment. The information provided will not be used as part of the data collection process. If participants are not eligible to participate, this information will be deleted (see Initial Screening Evaluation).

Once the initial Screening Evaluation has been received, the Principal Investigator (PI), Dr. Luis Columna, or his graduate and/or undergraduate students will contact participants to confirm that they have received the application. During this phone call, the study team will explain in more detail the purpose of the program, time commitment, potential risk, benefits, and answer any questions about the study.

The following steps describe the structure of the intervention (activities):

1. Parents in both groups will be asked to complete a Qualtrics survey (includes questions from Parenting Stress Index, TOPSE, DCDQ, and ABAS-3) inquiring about demographic information and or child's disability. This qualtrics survey will be embedded in the Fit Families App. *Note: The Fit Families app, which was developed by the study team using the Glide app. In this app, parents will receive a secured qualtrics link that will allow them to complete the surveys. The Fit Families App will not collect the data. However, it will be the mechanism to distribute the qualtrics surveys to the participants.
2. After the completion of the questionnaires, participants will be randomly assigned to one of two groups (e.g., intervention group or Wait-list control group). Group assignment will occur once pre-survey data has been collected. Each family will be notified via email or phone which group they have been assigned (e.g., Intervention or control group) within one week of the initial survey. The intervention group will be provided with the dates of the intervention workshop and mailed a set of physical activity equipment to use for practicing the skills outlined in the workshop. Similar approaches have been used in previous Fit Families program.

   * Participants in the intervention group will be offered four one-day group workshops (2-3 hours each) covering topics of 1) Sensory Integration, 2) Communication, 3) Physical activity, and 4) Sports. These workshops will be offered online via Zoom and will be video recorded. In addition to the workshops, the intervention group will receive information (activity booklets via the Fit Families App) and physical education (physical activity)-related equipment, which will be mailed to them. The activities discussed in the workshops are very similar to activities children will do during their physical education classes. During each workshop, parents will attend an online seminar and learn techniques and routines integrating the workshop topic into experiences. While attending the workshops, parents can ask questions using the chat feature of zoom or provided the opportunity to unmute themselves and ask questions to the speakers. The parents will also be able to show or send the study team videos/photos of them doing the activities with their child (which the research team will keep for research purposes if participant consents) so they can obtain feedback on their practice. The study team will provide a break in between for the participants. At the end of the workshop parents will be instructed to practice the skills they learned with their child for the next 3 weeks (for at least 3 hrs per week)

Zoom requires that users download an application to their computer or devices. The online portions of the workshop program will be either pre-recorded or distributed live to each family (depending on conversations with the Help Desk). Families will need to have access to internet services either through their phones or personal computers or devices. Note: To the investigator's knowledge, these families have already access to the internet or mobile technology because, in order to participate in the study, they are required to complete an online application. The online session will not include the practice component in which parents practice the skills learned with their children. In turn, the study team will ask families to share a video via box of them with their children practicing the skills. Each family will receive the equipment related to the workshop 2 days prior to the workshop. Staff from the Department of Kinesiology, in coordination with Dr. Columna or his graduate and undergraduate students, will mail the equipment to each family to the families in Wisconsin. The equipment to the families in Upstate New York, will be mailed by staff personnel from Syracuse University. The personnel at Syracuse will not have access to the identifiable data collected on participants. The duration of the online workshop will be approximately 2 and a half hours). Breaks will be provided as requested by the participants.

Participants in the intervention group will then be contacted by members of the research team on a weekly basis (during the length of the program) by text, or via email (depending on parental preferences) to encourage participation and usage of the games and activities provided.

At the culmination of the program, participants in the intervention group will be invited to participate in a focus group (via zoom) with members of the research team to explore their perception regarding communication strategies, patterns of physical recreation, perceived benefits, and constraints (see attached interview questions) and the duration of the focus group will be between 45 to 90 minutes. Breaks will be provided if necessary or if requested. The focus groups will also be video recorded.

• The wait-list home-based group will serve as the control group (during intervention). This group will be instructed to continue their typical routines and activities for the duration of the 12-week intervention. At the end of the 12 weeks, they will be asked to complete the post-test surveys (same as questionnaires completed prior to randomization). Their participation in the research will be complete at this time. However, because the intervention has been shown to potentially benefit families, immediately following the post-test, participants in the wait-list home-based group will be offered the chance to complete the home-based intervention program (e.g., receiving the same intervention protocol and materials (physical education equipment and lesson plans/workbook) as described for the intervention group). No data will be collected for research from them during this time

ELIGIBILITY:
Inclusion Criteria:

* Parents (one per family) of children with developmental and intellectual disabilities ages 4 to 11 will be included. Because this study is focused on families (parents) of children with developmental and intellectual disabilities, in order to participate, developmental and intellectual disabilities must be the primary disability. Children could have other disabilities besides developmental and intellectual disabilities, but developmental and intellectual disabilities must be their primary disability. Diagnostic severity of developmental and intellectual disabilities will not be a factor in recruitment. Recruitment will be based on diagnosis and the ability to participate in the program activities. Children must be ambulatory and able to follow verbal or picture directions with support. Children with significant communication needs will still be considered for the study. For adults (parents of children with developmental and intellectual disabilities) there will not be an age restriction. In addition, parents should be ambulatory and not have any restrictions to do physical activity. Lastly, because this study is focused on the States of Wisconsin and New York, participants need to reside either in the State of Wisconsin or in the State of New York, particularly upstate New York.

Note: While the children will be benefiting from this program, participants in this study will be the parents

Exclusion Criteria:

* Children with developmental and intellectual disabilities younger than 4 years old and older than 11 years old will be excluded from this research study. Because this study is focused on families (parents) of children with developmental and intellectual disabilities, parents of children with other primary disabilities, or parents who do not have children with developmental and intellectual disabilities will be excluded. Participants cannot exhibit aggressive behavior. Children who are non-ambulatory or participants (children) with significant behavioral or sensory impairments will also be excluded based on application information, including existing behavior intervention plans and existing school information. Participants who are not residents of the States of New York or Wisconsin will not be able to participate in this study.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
Change in Parenting Stress Index (PSI)- Short form | Baseline, 3 week post intervention (15 weeks)
  The Parenting Stress Index (PSI)- short form is used to measure the relative stress in the parent-child relationship. Parents complete the PSI Short Form test sheet including basic demographic information on the top of the questionnaire first. For most items, parents should respond by circling SA (strongly agree), A (agree), NS (not sure), D (disagree), SD (strongly disagree). Higher raw scores indicate higher levels of stress. Percentile scores that fall between 15 and 80 are considered typical.
Change in Adaptive Behavior Assessment System (ABAS-3) | Baseline, 3 week post intervention (15 weeks)
  To evaluate adaptive behavior skills of the child. The ABAS-3 covers three broad adaptive domains: Conceptual, Social, and Practical. Within these domains, it assesses 11 adaptive skill areas (each form assesses 9 or 10 skill areas based on age range). Items focus on practical, everyday activities required to function, meet environmental demands, care for oneself, and interact with others effectively and independently. On a four-point response scale, raters indicate whether the individual can perform each activity, and if so, how frequently they perform it when needed. The ratings for each skill are converted into a score from 1 to 19 with a higher score indicative of higher adaptive behavior skills.
DCDQ: Developmental Coordination Disorder Questionnaire | Baseline, 3 week post intervention (15 weeks)
  The Developmental Coordination Questionnaire (DCDQ) is a parent report measure developed to assist in the identification of Developmental Coordination Disorder (DCD) in children. Parents are asked to compare their child's motor performance to that of his/her peers using a 5 point Likert scale. Most of the motor skills that this questionnaire asks about are things that a child does with his or her hands, or while moving. The scale ranges from 1 (not at all like your child) to 5 (extremely like your child).
TOPSE: Tool to measure Parenting Self-Efficacy | Baseline, 3 week post intervention (15 weeks)
  TOPSE: Tool to measure Parenting Self-Efficacy is used to measure play and enjoyment. The scale ranges from 0 (completely disagree) to 10 (completely agree). On a ten-point response scale, raters indicate how much they agree with each statement

CONTACTS AND LOCATIONS:
Overall Officials: Luis Columna, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin- Madison, Madison, Wisconsin, United States